CLINICAL TRIAL: NCT03338218
Title: Pragmatic, Prospective, Randomized, Controlled, Double-blind, Multi-centre, Multinational Study on the Safety and Efficacy of a 6% Hydroxyethyl Starch (HES) Solution Versus an Electrolyte Solution in Trauma Patients
Brief Title: Safety and Efficacy of a 6% Hydroxyethyl Starch (HES) Solution Versus an Electrolyte Solution in Trauma Patients
Acronym: TETHYS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Collaborators: B. Braun Melsungen AG (Industry); European Society of Anaesthesiology and Intensive Care (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HC-G-H-1505; HE06-021-CP4 (Other: Fresenius Kabi)
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Hypovolemia Due to Acute Blood Loss
Keywords: Hydroxyethyl starch; HES; HES 130
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Volulyte 6% (Experimental): Volulyte 6% solution for infusion
  Interventions: Drug: Volulyte 6%
- Ionolyte (Active Comparator): Ionolyte solution for infusion
  Interventions: Drug: Ionolyte

INTERVENTIONS:
Drug: Volulyte 6% — Solution for infusion
  Other Names: Hydroxyethyl starch 130
  Arms: Volulyte 6%
Drug: Ionolyte — Solution for infusion
  Other Names: Ionolyte Electrolyte Solution
  Arms: Ionolyte

SUMMARY:
The aim of the study is to investigate the safety of a 6% hydroxyethyl starch (HES) solution (Volulyte 6%) versus an electrolyte solution (Ionolyte) in trauma patients.

ELIGIBILITY:
Inclusion:

* Male or female adult patients ≥18 years of age. Women of child bearing potential must test negative on standard pregnancy test (urine or serum) (as soon as possible during emergency care)
* Patients with blunt or penetrating trauma suffering from estimated blood loss of ≥ 500 ml
* Initial surgery deemed necessary within 24 hrs after trauma
* Deferred signed written informed consent form or as locally required
* No signs of intracranial or cerebral hemorrhage
* Administration of less than 15 ml/kg body weight colloid between trauma injury and hospital admission.

Exclusion:

* Hypersensitivity to the active substances or to any of the other excipients of the Investigational Products
* Body weight ≥ 140 kg
* Patients expected to die within 24h after traumatic injury
* Sepsis
* Burns
* Renal impairment (AKIN stage ≥ 1 or chronic) or acute and/or chronic Renal Replacement Therapy
* Critically ill patients (typically admitted to the intensive care unit)
* Hyperhydration
* Pulmonary edema
* Dehydration
* Hyperkalemia
* Severe hypernatremia
* Severe hyperchloremia
* Severely impaired hepatic function
* Congestive heart failure
* Severe coagulopathy
* Organ transplant patients
* Metabolic alkalosis
* Simultaneous participation in another interventional clinical trial (drugs or medical devices studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2019-02-23 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of 90 day mortality and 90 day renal failure defined as biomarker increase as defined by AKIN stage 2 or RIFLE injury stage or need for RRT at any time during the first 3 months. | 90 days

SECONDARY OUTCOMES:
Serum creatinine | 7 days post-trauma
Serum creatinine-based estimated glomerular filtration rate | 7 days post-trauma
Cystatin-C | 3 days post-trauma
Cystatin-C-based mean estimated glomerular filtration rate | 3 days post-trauma
AKIN stages | 7 days post-trauma
Highest AKIN stage reached on each day during the first week | 7 days post-trauma
RIFLE stages | 7 days post-trauma
Urine output (if available) | 7 days post-trauma
Days on Renal Replacement Therapy | 90 days after randomization
Patients on Renal Replacement Therapy | 90 days after randomization
Platelet count | 3 days post-trauma
International normalized ratio | 3 days post-trauma
Activated partial thromboplastin time | 3 days post-trauma
Adverse Events | 90 days after randomization
Mortality | 90 days after randomization
Length of Stay in ICU/hospital | 90 days after randomization
C-reactive protein | 3 days post-trauma
Hours on mechanical ventilation | 7 days post-trauma
Total volume of administered investigational products | until 24 hours after investigational product treatment start
Fluid balance | 7 days post-trauma
  Sum of volume of all intravenous medication (including investigational product and blood products) minus sum of volume of urine output (if available), drainage and estimated due to surgeries and trauma
Heart rate | 7 days post-trauma
Temperature | 7 days post-trauma
Mean arterial pressure | 7 days post-trauma
Systolic arterial blood pressure | 7 days post-trauma
Diastolic arterial blood pressure | 7 days post-trauma
Central venous pressure (if available) | 7 days post-trauma
Partial pressure of carbon dioxide | 3 days post-trauma
Partial pressure of oxygen | 3 days post-trauma
Bicarbonate | 3 days post-trauma
Arterial oxygen saturation | 3 days post-trauma
Hemoglobin | 3 days post-trauma
Hematocrit | 3 days post-trauma
pH | 3 days post-trauma
Base excess | 3 days post-trauma
Lactate | 3 days post-trauma
Central venous oxygen saturation (if available) | 3 days post-trauma
Serum sodium | 3 days post-trauma
Serum potassium | 3 days post-trauma
Serum calcium | 3 days post-trauma
Serum chloride | 3 days post-trauma

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang F. Buhre, Prof. Dr. med., Study Chair — Department of Anesthesiology and Pain Management, Maastricht University, The Netherlands
Locations (22):
- Ziekenhuis Oost-Limburg-ZOL, Genk, Belgium
- Czechia (2):
  - Fakultni nemocnice Brno, Brno
  - Military University Hospital, Prague
- France (2):
  - CHRU Nancy - Hôpital Central, Nancy
  - Hôpital de Hautepierre, Strasbourg
- Germany (4):
  - Universitätsklinikum Aachen, Aachen
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Frankfurt, Frankfurt
  - University Hospital Schleswig-Holstein Campus Kiel, Kiel
- Netherlands (2):
  - Academic Medical Center (AMC) Anesthesiology, Amsterdam
  - University Medical Center (UMC) Maastricht, Maastricht
- South Africa (8):
  - Groote Schuur Hospital, Cape Town
  - Gama Research Centre Emergency Department, Leratong Hospital, Germiston
  - Gama Research Centre, Germiston
  - Chris Hani Baragwanath Hospital, Johannesburg
  - Trident Clinical, Homestead Medical Centre, Kimberley
  - Steve Biko Academic Hospital, Pretoria
  - FCRN Clinical Trials Centre, Vereeniging
  - Clinical Projects Research SA, Worcester
- Spain (3):
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Clinico Universitario, Valencia
  - Hospital Universitari i Politecnic la Fe, Valencia

REFERENCES:
- [Derived] Palma CD, Mamba M, Geldenhuys J, Fadahun O, Rossaint R, Zacharowski K, Brand M, Diaz-Cambronero O, Belda J, Westphal M, Brauer U, Dormann D, Dehnhardt T, Hernandez-Gonzalez M, Schmier S, de Korte D, Plani F, Buhre W. PragmaTic, prospEctive, randomized, controlled, double-blind, mulTi-centre, multinational study on the safety and efficacy of a 6% HydroxYethyl Starch (HES) solution versus an electrolyte solution in trauma patients: study protocol for the TETHYS study. Trials. 2022 Jun 2;23(1):456. doi: 10.1186/s13063-022-06390-x. PMID 35655234
- [Derived] Chappell D, Jacob M. Should hydroxyethyl starch be banned? Lancet. 2018 Jul 14;392(10142):118. doi: 10.1016/S0140-6736(18)31174-7. No abstract available. PMID 30017128